CLINICAL TRIAL: NCT05142891
Title: Incidence of Actue Kidney Injury in Patients Treated With Amoxicillin and Cloxacillin Combination Therapy
Brief Title: Renal Tolerance of Amoxicillin and Cloxacillin Combination
Acronym: Amox-Cloxa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8411
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Endocarditis; Acute Kidney Injury
Keywords: Endocarditis; Acute kidney injury; Amoxicillin; Cloxacillin
MeSH Terms: conditions — Endocarditis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
2015 European Society of Cardiology Guidelines have proposed the combination of Ampicillin and Cloxacillin for initial empirical treatment of infective endocarditis in acute severely ill patients (before pathogen identiﬁcation). Yet this combination has never been studied in clinical trials. High dose penicillin treatments are associated with a risk of nephrotoxicity.

The investigator's primary purpose is to describe patients treated with high dose Amoxicillin and Cloxacillin combination and to evaluate its renal tolerance.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Hospitalized at the Strasbourg University Hospital and treated concomitantly with Amoxicillin IV and Cloxacillin IV for ≥48 hours between January 1, 2016 and December 31, 2020.
* Patient not having expressed his opposition, after information, to the reuse of his data for scientific research purposes.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient hospitalized at the Strasbourg University Hospital and treated concomitantly with Amoxicillin IV and Cloxacillin IV for ≥48 hours between January 1, 2016 and December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Description of patients treated with dual IV therapy combining cloxacillin and amoxicillin in high doses at Strasbourg University Hospital | Files analysed retrospectively from January 01, 2016 to December 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Yvon RUCH, MD, Principal Investigator — Service de maladies infectieuses et tropicales - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de maladies infectieuses et tropicales - Hôpitaux Universitaires de Strasbourg, Strasbourg, France